CLINICAL TRIAL: NCT01976572
Title: A Randomised, Open-Label, Drug-Drug Interaction Study to Evaluate the Effect of Colestilan on the Pharmacokinetics of Single Oral Doses of Candesartan Cilexetil in Healthy Subjects
Brief Title: Drug-Drug Interaction Study to Evaluate the Effect of Colestilan on the Pharmacokinetics of Single Doses of Candesartan Cilexetil in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MCI-196-E17
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Hyperphosphatemia; Chronic Kidney Disease
Keywords: CKD Stage V; dialysis
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic | interventions — cholebine; candesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Candesartan alone (Placebo Comparator): Single dose of 16 mg candesartan was administered orally on Day 1.
  Interventions: Drug: candesartan
- T0hr (Active Comparator): Colestilan was administered orally 5 g t.i.d (total dose 15 g/day) in the fed state immediately after meals from Day 3 to Day 24 and single dose of 16 mg candesartan was administered orally on Day 7, 13 and 19 at 1 of 3 dosing time-points relative to the first daily dose of 5 g colestilan t.i.d. T-0 of 3 dosing time-points means the single dose of candesartan was administered at the same time relative to the first daily dose of colestilan.
  Interventions: Drug: colestilan; Drug: candesartan
- T-1hr (Active Comparator): Colestilan was administered orally 5 g t.i.d (total dose 15 g/day) in the fed state immediately after meals from Day 3 to Day 24 and single dose of 16 mg candesartan was administered orally on Day 7, 13 and 19 at 1 of 3 dosing time-points relative to the first daily dose of 5 g colestilan t.i.d. T-1 of 3 dosing time-points means the single dose of candesartan was administered at 1 hour before relative to the first daily dose of colestilan.
  Interventions: Drug: colestilan; Drug: candesartan
- T+3hr (Active Comparator): Colestilan was administered orally 5 g t.i.d (total dose 15 g/day) in the fed state immediately after meals from Day 3 to Day 24 and single dose of 16 mg candesartan was administered orally on Day 7, 13 and 19 at 1 of 3 dosing time-points relative to the first daily dose of 5 g colestilan t.i.d. T+3 of 3 dosing time-points means the single dose of candesartan was administered at 3 hour after relative to the first daily dose of colestilan.
  Interventions: Drug: colestilan; Drug: candesartan

INTERVENTIONS:
Drug: colestilan
  Other Names: BindRen
  Arms: T+3hr; T-1hr; T0hr
Drug: candesartan

SUMMARY:
The primary objective is to assess the effects of colestilan on the pharmacokinetic profile of candesartan cilexetil when administered at the same time as, 1 hour before, and 3 hours after the first daily dose of colestilan administered at doses of 5 g three times daily compared to administration of candesartan cilexetil alone, in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent to participate in this study, after reading the participant information sheet and informed consent form (ICF), and after having the opportunity to discuss the study with the Investigator or designee.
* Caucasian male subjects aged 18 to 50 years inclusive.
* A body mass index (BMI) between 18.0 and 32.0 kg/m2, both inclusive.
* Healthy subjects, free from any clinically significant illness or disease as determined by their medical history, physical examination, electrocardiogram (ECG), vital signs, biochemistry, haematology, coagulation, urinalysis, and serology.
* Male subjects, and their partners, agree to use contraception throughout the study duration. Male subjects must use 1 barrier method of contraception and spermicide during the trial, and for 3 months after the last dose of study drug. Male subjects with female partners of child-bearing potential must also agree to use an additional highly effective method of contraception. They must use a condom, and their female partners must use an additional method of contraception (such as cap or diaphragm), unless the subject or his partner has been sterilised, in which case, male subjects must use a condom and spermicide.

Exclusion Criteria:

* Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration, as determined by the Investigator based on abnormal medical history, physical findings, or laboratory values at Screening or Baseline.
* Unable to swallow colestilan tablets, current and/or history of dysphagia.
* Current or any history of any of the following gastrointestinal (GI) diseases: intestinal obstruction, chronic or severe constipation, subileus, ileus, intestinal stenosis, intestinal diverticulosis and/or diverticulitis, colitis, GI ulcers, recent major GI surgery, peritonitis, GI bleeding, gastritis, haemorrhoids, or any other severe GI disease.
* Current or any history of biliary obstruction, cholestasis, or severe hepatic impairment.
* Current or history of seizure disorders.
* Current or history of Vitamin K deficiency.
* Subjects who have any clinically significant allergic disease (excluding non-active hayfever) as determined by the Investigator.
* Current or recent history (in the last 2 years) of abuse or addiction (tobacco, alcohol, drugs or substances), or weekly alcohol intake of more than 21 units, or a positive alcohol breath test or urine drug screen at Screening or Baseline. One unit is equivalent to a ½ pint (280 mL) of beer, 1 measure (25 mL) of spirits or 1 small glass (125 mL) of wine.
* Treatment with any drugs or herbal or dietary supplements known to be inhibitors of cytochrome P450 (CYP) 3A4, CYP2C9 or P-glycoprotein, 7 days before dosing and inducers of CYP3A4, CYP2C9, or P-glycoprotein 14 days before dosing.
* Treatment with H2 antagonist and/or proton pump inhibitors, during 4 weeks before dosing.
* Subjects with a history of hypotension or hyperkalaemia, or a postural drop of systolic blood pressure ≥20 mmHg at Screening.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, Dr, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, Springfield House Hyde Street, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Covance from 14th October 2013.
Groups:
- Treatment A: On Day 1, a single dose of candesartan (16 mg) was administered. On Day 7, the first daily dose of colestilan (5 g) and candesartan were administered together (T0). On Day 13, candesartan was administered at 1 hour before (T-1) the first daily dose of colestilan, and on Day 19 at 3 hours after (T+3) the first daily dose of colestilan.
- Treatment B: On Day 1, a single dose of candesartan (16 mg) was administered. On Day 7, candesartan was administered at 1 hour before (T-1) the first daily dose of colestilan. On Day 13, candesartan was administered at 3 hours after (T+3) the first daily dose of colestilan, and on Day 19, the first daily dose of colestilan and candesartan were administered together (T0).
- Treatment C: On Day 1, a single dose of candesartan (16 mg) was administered. On Day 7, candesartan was administered at 3 hours after (T+3) the first daily dose of colestilan. On Day 13, the first daily dose of colestilan and candesartan was administered together (T0), and on Day 19 candesartan was administered at 1 hour before (T-1) the first daily dose of colestilan.
Period: Overall Study
Arm/Group | Treatment A | Treatment B | Treatment C
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: AUC0-t of Candesartan
Description: Area under the plasma concentration-time curve from time zero up to the last quantifiable time-point
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: PK Population: All subjects who receive at least one dose of candesartan and have sufficient interpretable PK data.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Candesartan Alone: Single dose of candesartan (16 mg) only
- T-1hr: Single dose of candesartan (16 mg) with colestilan (5 g three times daily) co-administration at 1 hour before
- T0hr: Single dose of candesartan (16 mg) with colestilan (5 g three times daily) co-administration at the same time
- T+3hr: Single dose of candesartan (16 mg) with colestilan (5 g three times daily) co-administration at 3 hour after
Arm/Group | Candesartan Alone | T-1hr | T0hr | T+3hr
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng*hr/mL | 1118 (249) | 826 (308) | 494 (127) | 759 (211)

2. Primary Outcome: Cmax of Candesartan
Description: Maximum observed plasma concentration
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, and 48 hours post-dose
Population: PK Population: All subjects who receive at least one dose of candesartan and have sufficient interpretable PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Candesartan Alone | T-1hr | T0hr | T+3hr
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng/mL | 106.7 (37.9) | 94.7 (58.3) | 42.8 (7.0) | 99.5 (36.9)

3. Secondary Outcome: Tmax
Description: Time of maximum observed plasma concentration
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, and 48 hours post-dose
Measure: Median (Full Range); unit: hr
Arm/Group | Candesartan Alone | T-1hr | T0hr | T+3hr
Number analyzed (Participants) | 18 | 18 | 18 | 18
hr | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 8.00] | 5.05 [3.00 to 5.12] | 2.05 [2.05 to 5.00]

4. Secondary Outcome: T1/2
Description: Apparent plasma terminal elimination half-life
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, and 48 hours post-dose
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Candesartan Alone | T-1hr | T0hr | T+3hr
Number analyzed (Participants) | 18 | 18 | 18 | 18
hr | 13.50 (3.31) | 9.61 (1.90) | 10.44 (2.18) | 10.01 (1.73)

ADVERSE EVENTS:
Time Frame: 24 days
Arm/Group | Candesartan Alone (Day 1 to 2) | Colestilan Alone (Day 3 to 6) | Candesartan Plus Colestilan (Day 7 to 24)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 5/18 | 10/18 | 11/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan Alone (Day 1 to 2) (N=18) | Colestilan Alone (Day 3 to 6) (N=18) | Candesartan Plus Colestilan (Day 7 to 24) (N=18)
Nausea (Gastrointestinal disorders) | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 2
Lethargy (Nervous system disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 2
Chest pain (General disorders) | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Eyelid skin dryness (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 1
Middle insomnia (Psychiatric disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other